CLINICAL TRIAL: NCT03558906
Title: Gingival Crevicular Fluid and Salivary HIF-1α, VEGF and TNF-α Levels in Different Periodontal Diseases
Brief Title: TNF-α/HIF-1α/VEGF Pathway in Periodontal Diseases
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Collaborators: Celal Bayar University (Other); Ege University (Other)
Responsible Party: Principal Investigator, Beral Afacan, Assistant Professor, Aydin Adnan Menderes University
Other Study IDs: bafacan357
Record Dates: First submitted 2018-05-23; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Periodontal Diseases
Keywords: Periodontal disease; Hypoxia; Cytokines; Gingival crevicular fluid; Saliva
MeSH Terms: conditions — Periodontal Diseases; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid, saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Aggressive Periodontitis: These individuals had minimum PD ≥6 mm and CAL ≥5 mm on eight or more teeth; at least three of these were other than central incisors or first molars. Radiographic alveolar bone loss was ≥30% of root length affecting at least three permanent teeth other than first molars and incisors. The severe destruction pattern was not commensurate with amount of plaque accumulation.
- Chronic periodontitis: These individuals had at least four non-adjacent teeth with sites with PD ≥6 mm and CAL ≥5 mm. They had also ≥50% alveolar bone loss in at least two quadrants that was commensurate with amount of plaque accumulation. BOP was >50% in the whole mouth.
- Gingivitis: Gingivitis patients exhibited no sites with CAL >2 mm and no detectable alveolar bone loss in the radiography. BOP was >50% in the whole mouth.
- Healthy: Periodontally healthy volunteers exhibited no sites with PD >3 mm and CAL >2 mm as well as no radiographic evidence of alveolar bone loss. BOP was <15% in the whole mouth.

SUMMARY:
This study aimed to investigate gingival crevicular fluid (GCF) and salivary hypoxia inducible factor-1 alpha (HIF-1α), vascular endothelial growth factor (VEGF) and tumor necrosis factor-alpha (TNF-α) levels in different periodontal diseases. A total of 87 individuals, 20 patients with generalized aggressive periodontitis, 20 with chronic periodontitis, 26 with gingivitis and 21 periodontally healthy individuals were included. Whole-mouth and site-specific clinical periodontal parameters including probing depth, clinical attachment level, bleeding on probing, gingival index and plaque index were recorded. GCF and salivary HIF-1α, VEGF and TNF-α levels were measured by enzyme-linked immunosorbent assay. Statistical analysis was performed by using non-parametric tests.

DETAILED DESCRIPTION:
Study Population and Clinical Examination

Eighty-seven participants were recruited for the study. Exclusion criteria were as follows: 1) systemic diseases that could affect the periodontium; 2) smoking; 3) current pregnancy or lactation; 4) nonsurgical/surgical periodontal treatment received for the past year; and 5) use of anti-inflammatory and antibiotic drugs within the past 6 months.

The full-mouth clinical periodontal examination included measurement of probing depth (PD), clinical attachment level (CAL), presence of bleeding on probing (BOP), gingival index (GI) and plaque index (PI) at 6 sites per tooth. Presence and extent of alveolar bone loss were assessed radiographically. Based on clinical and radiographic diagnostic criteria proposed by 1999 International Workshop for a Classification of Periodontal Diseases and Conditions, the participants were categorized into four groups.

I. Generalized aggressive periodontitis (GAgP) group (n=20). These individuals had minimum PD ≥6 mm and CAL ≥5 mm on eight or more teeth; at least three of these were other than central incisors or first molars. Radiographic alveolar bone loss was ≥30% of root length affecting at least three permanent teeth other than first molars and incisors. The severe destruction pattern was not commensurate with amount of plaque accumulation or other local risk factors for a given age.

II. Chronic periodontitis (CP) group (n=20). These individuals had at least four non-adjacent teeth with sites with PD ≥6 mm and CAL ≥5 mm. They had also ≥50% alveolar bone loss in at least two quadrants that was commensurate with amount of plaque accumulation. BOP was >50% in the whole mouth.

III. Gingivitis group (n=26). These individuals had varying degrees of gingival inflammation. They exhibited no sites with CAL >2 mm and no detectable alveolar bone loss in the radiography. BOP was >50% in the whole mouth.

IV. Healthy group (n=21). These periodontally healthy volunteers exhibited no sites with PD >3 mm and CAL >2 mm as well as no radiographic evidence of alveolar bone loss. BOP was <15% in the whole mouth.

Saliva sampling

Whole unstimulated saliva samples were collected. Each participant was asked first to rinse the mouth completely with tap water for 2 minutes, wait for 10 minutes, and then expectorate into sterile polypropylene tube for 5 minutes.

Gingival crevicular fluid (GCF) sampling

Standardized filter paper strips were used for GCF sampling. Two GCF samples were taken from the buccal aspects of two non-adjacent interproximal sites of each individual. In patients with periodontitis, GCF were sampled from two sites exhibiting PD ≥6 mm and CAL ≥5 mm. GCF samples of gingivitis patients were obtained from the sites that exhibit BOP but no clinical attachment loss. In the healthy group, GCF samples were collected the sites exhibiting PD <3 mm without BOP and clinical attachment loss.

Measurement of hypoxia inducible factor-1 alpha (HIF-1α), vascular endothelial growth factor (VEGF) and tumor necrosis factor-alpha (TNF-α) Levels in GCF and Saliva Samples

HIF-1α, VEGF and TNF-α levels in GCF and saliva samples were measured by the enzyme-linked immunosorbent assay (ELISA) using commercial kits according to the manufacturer's guidelines.

Statistical Analysis

All data analyses were performed using a statistical software package. Comparisons of clinical and biochemical parameters between the study groups were performed using the Kruskal-Wallis test.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy individuals
2. Non-smoker individuals

Exclusion Criteria:

1. Current pregnancy or lactation
2. Nonsurgical/surgical periodontal treatment received for the past year
3. Use of anti-inflammatory and antibiotic drugs within the past 6 months.

Ages: 27 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All consecutive individuals were recruited from the Department of Periodontology, School of Dentistry, Adnan Menderes University, Aydın.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-03-02 (Actual); Study Completion 2016-12-26 (Actual)

PRIMARY OUTCOMES:
Gingival crevicular fluid HIF-1α levels | A day after clinical periodontal examination
  pg

SECONDARY OUTCOMES:
Salivary HIF-1α levels | A day after clinical periodontal examination
  pg/ml
Gingival crevicular fluid VEGF levels | A day after clinical periodontal examination
  ng
Salivary VEGF levels | A day after clinical periodontal examination
  ng/l

REFERENCES:
- [Derived] Afacan B, Ozturk VO, Pasali C, Bozkurt E, Kose T, Emingil G. Gingival crevicular fluid and salivary HIF-1alpha, VEGF, and TNF-alpha levels in periodontal health and disease. J Periodontol. 2019 Jul;90(7):788-797. doi: 10.1002/JPER.18-0412. Epub 2018 Dec 11. PMID 30536725